CLINICAL TRIAL: NCT02114541
Title: Global Observational Study to Evaluate the Correlation Between Coronary and Carotid Atherosclerotic Disease (CAD) and Links With Clinical Outcomes
Brief Title: Correlation Between Coronary and Carotid Atherosclerotic Disease and Links With Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CAIN-003_MHICC-31052012
Record Dates: First submitted 2013-07-18; First posted 2014-04-15 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Vascular Disease
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The relationship of the natural history of atherosclerosis between different vascular beds has not been well characterized. Determination and comparison of the relative rates of progression and extents of atherosclerosis in the coronary and carotid arterial trees may have major impacts on clinical research and clinical practice. Correlation between findings in the carotid and coronary circulations is an important scientific and clinical topic to address. Results from a well design study incorporating imaging technologies that currently represent the gold standards for the assessment of coronary and carotid artery plaque burden, will have potentially impact on clinical research and clinical practice.

DETAILED DESCRIPTION:
The CAIN-003 study was a prospective observational multi-center imaging study of subjects scheduled for clinically-indicated coronary angiography. CAIN-003 provided for the collection of baseline coronary angiography and IVUS imaging data along with baseline carotid ultrasound imaging. CAIN-003 study participants underwent follow-up coronary and carotid imaging at 2-years, and were then contacted by phone on an annual basis for an additional 3 years for the collection of cardiovascular and cerebrovascular clinical endpoints.

MHICC-31052012 was a prospective, observational, multi-center study of subjects who had successfully undergone baseline imaging in the dal-PLAQUE 2 study (A multicenter, double-blind, randomized, placebo-controlled study, evaluating the effect of treatment with dalcetrapib 600 mg on atherosclerosis disease). The dal-PLAQUE 2 study, which provided for the collection of baseline and 2-year follow-up coronary angiography, coronary IVUS and carotid ultrasound imaging data, was terminated by the sponsor prior to completion due to the discontinuation of the dalcetrapib drug development program. The MHICC-31052012 study allowed for the collection of follow-up imaging and clinical endpoint data from subjects who had successfully undergone baseline IVUS imaging in dal-PLAQUE 2.

Data from CAIN-003 and MHICC-31052012 was pooled to support the objective of determining the correlation and clinical relevance of these imaging endpoints.

The objectives of the CAIN-003 and MHICC-31052012 study were:

* To compare the extent of atherosclerosis present in the coronary vasculature with the extent of atherosclerosis present in the carotid vasculature at a single point in time.
* To compare the associations of atherosclerosis burden with coronary risk factors in the coronary arteries and carotid arteries, in multivariable regression.
* To compare the rate of atherosclerosis progression or regression in the coronary vasculature with the rate of atherosclerosis progression or regression in the carotid vasculature over a 2-year period.
* To determine the correlation between imaging biomarkers and cardiovascular outcomes over a 5-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients over the age of 18 years.
2. Patients scheduled for clinically indicated coronary angiography and possible ad hoc percutaneous coronary intervention (PCI) will be evaluated before their scheduled procedure.
3. Written informed consent (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) obtained prior to any study specific procedures.
4. Patients considered to be stable at enrollment (at the discretion of the investigator) are eligible provided they meet all other entry criteria.
5. Angiographic inclusion criteria:

   * Entire Coronary Circulation: The patient must have angiographic evidence of coronary artery disease as defined by at least one lesion in any of the three major native coronary arteries that has >20% reduction in lumen diameter by angiographic visual estimation or prior history of PCI. This vessel does not need to be the target coronary artery for IVUS. Any vessel with previous PCI may not be used as the target coronary artery.
   * Left Main Coronary Artery: The patient must not have > 50% reduction in lumen diameter by visual angiographic estimation.
   * Target Coronary Artery: Patient will be required to have one "target" coronary artery for IVUS that has not undergone prior PCI, that is not a candidate to undergo PCI presently or in the next 24 months, and that has not been the cause of a recent myocardial infarction. The proximal 4 cm of the "target" artery in which

IVUS examination will be performed at baseline:

* Must have a diameter stenosis < 50% lumen diameter by visual assessment of the angiogram;
* Must have a reference diameter > 2.5 mm;
* Must be free of filling defects suggestive of thrombus;
* Must not present any anatomical characteristic (such as but not limited to severe tortuosity or calcification) that would impede IVUS interrogation at baseline or follow-up
* Note: a lesion of up to 60% stenosis is permitted, distal to the target segment. A side branch of the target coronary artery for IVUS may not be a target for PCI.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Women of childbearing potential (women who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who refuse to undergo a urine or serum pregnancy test immediately prior to baseline and repeat imaging evaluations The urine or serum pregnancy test must be negative prior to imaging evaluations.
2. Previous coronary artery bypass graft (CABG) surgery or probable need for CABG in the next 24 months.
3. Patients who have symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Class III or IV) at baseline.
4. Patients with clinically significant valvular heart disease likely to require surgical repair or replacement during the treatment period of the study
5. Any clinically significant medical condition or presence of any laboratory abnormality that is considered by the investigator to be clinically important and could interfere with the conduct of the study.
6. The presence of severe liver disease as defined by the presence of cirrhosis, chronic active hepatitis, or chronic jaundice with hyperbilirubinemia,
7. Patients with eGFR < 45 ml/min prior to baseline imaging procedures, or with nephrotic syndrome
8. Patients with a life expectancy less than 2 years.
9. History of malignancy (except for curatively treated basal cell or squamous cell carcinoma of the skin) during the 3 years prior to the screening.
10. Unable or unwilling to comply with protocol requirements, or deemed by the investigator to be unfit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who were scheduled for clinically-indicated coronary angiography and undergone baseline coronary angiography and IVUS imaging data along with baseline carotid ultrasound imaging.
Sampling Method: Non-Probability Sample
Enrollment: 1339 (Actual)
Dates: Start 2010-02-03 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Nominal change at follow-up from baseline in percent atheroma volume (PAV) obtained using intravascular ultrasound (IVUS) | Participants will have a baseline IVUS and a two year follow-up IVUS
  This endpoint will be the nominal change at follow-up from baseline in percent atheroma volume computed by dividing plaque volume by external elastic membrane volume and then multiplying by 100 at both time points, baseline and 2 year follow-up.

SECONDARY OUTCOMES:
plaque volume in target coronary artery | change at 2 year follow-up from baseline
  This secondary IVUS endpoint will include the nominal change in plaque volume in the target coronary artery, as well as the percent (relative) change in plaque volume.
change in plaque volume in the 5-mm sub-segment of target coronary artery | change at 2 year follow-up from baseline
  change in plaque volume in the 5-mm sub-segment with the greatest disease burden at baseline, and change in plaque volume in the 5-mm sub-segment with the smallest plaque area at baseline.
Total vessel volume in the target coronary artery | change at final 2 year follow-up from baseline
  Total vessel volume for all anatomically comparable slices in the 30-mm target coronary artery segment and the change in plaque characterization indices.
change in coronary score assessed by quantitative coronary angiography | change at final 2 year follow-up from baseline
  Evaluation of change in coronary score assessed by quantitative coronary angiography and defined as the per-patient mean of the minimal lumen diameter for all lesions measured. As well evaluation of the cumulative coronary stenosis score (calculated by adding all percent diameter stenoses in standard international units).
nominal change in carotid IMT(CIMT) | change at final 2 year follow-up from baseline
  This secondary endpoint will be obtained using 2D B-mode carotid ultrasound and will be the nominal change at final follow-up from baseline in carotid IMT(CIMT), where CIMT is computed as the per scan average of the mean IMT values of carotid segments.

OTHER OUTCOMES:
clinical endpoints | up to five year follow-up
  Clinical endpoints: death, coronary heart disease, resuscitated cardiac arrest, non-fatal myocardial infarction, stroke, hospitalization for documented acute coronary syndrome (ECG abnormalities without biomarkers), coronary revascularization procedure and carotid artery surgery or angioplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, M.D, Principal Investigator — Montreal Heart Institute
Locations (69):
- United States (16):
  - University of southern California, Los Angeles, California
  - Los Angeles Biomedical Research Institute at Harbor, Torrance, California
  - Jim Moran Heart and Vascular Research Institute, Holy Cross Hospital, Fort Lauderdale, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Florida Cardiovascular Research, Tampa, Florida
  - Emory University VA Medical Center, Decatur, Georgia
  - Norton Heart Specialist Springs, Louisville, Kentucky
  - John Hopkins University Office Capitol Region Research-CAPRES, Columbia, Maryland
  - CV Research at MidMichigan Medical Center Midland, Midland, Michigan
  - Mercy Health Partners, Muskegon, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - The Valley Hospital, Ridgewood, New Jersey
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - University of Toledo Medical Center, Toledo, Ohio
  - Parkway Cardiology associates, Oak Ridge, Tennessee
  - Dalla VAMC, Dallas, Texas
- Canada (40):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Mazankowski Alberta Heart Institute University Of Alberta Hospital ABACUS, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Interventional Cardiology Research, St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation (Office)/Royal Jubilee Hospital, Victoria, British Columbia
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II - Health Sciences Centre, Halifax, Nova Scotia
  - Cambridge Cardiac Care, Cambridge, Ontario
  - McMaster Clinic Hamilton General Hospital, Hamilton, Ontario
  - KMH Cardiology & Diagnostics Centre, Kitchener, Ontario
  - University Hospital/LHSC, London, Ontario
  - KMH Cardiology & Diagnostics Centre, Mississauga, Ontario
  - York PCI Research, Newmarket, Ontario
  - Heart Care Research, Oshawa, Ontario
  - Ottawa Civic Hospital / University of Ottawa Heart Institute, Ottawa, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Complexe Hospitalier de la Sagamie, Chicoutimi, Quebec
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - CSSS-Hopital de Gatineau, secteur Hull, Gatineau, Quebec
  - Q & T Research, Gatineau, Quebec
  - Viacar Recherche Clinique, Greenfield Park, Quebec
  - Cite de la Sante, Laval, Quebec
  - CDRC Rive Sud, Longueuil, Quebec
  - Foothills Medical Centre, Longueuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM - Hopital Hotel-Dieu, Montreal, Quebec
  - CUSM Montreal General Hospital, Montreal, Quebec
  - Hopital Sacré-Cœur de Montreal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Centre Hospitalier Régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - Centre de santé et des services sociaux de Beauce, Saint-Georges, Quebec
  - St-Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - Sunnybrook Health Science Center, Toronto, Quebec
  - Centre de santé et de services sociaux de Trois-Rivières, Trois-Rivières, Quebec
  - CSSS Vallée de l'Or, Val-d'Or, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Foothills Medical Centre, Calgary
- Germany (4):
  - Universitatsklinikum Aachen, Aachen
  - Klinikum Darmstadt, Darmstadt
  - Universitat Heidelberg, Heidelberg
  - Universitatsklinikum Ulm, Ulm
- Poland (8):
  - Wojewodzki Szpital, Elblag
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Oddzial Kliniczny Choroby, Krakow
  - Samodzielny Publiczny, Lublin
  - Szpital Kliniczny, Poznan
  - Klinika Kardiologii, Warsaw
  - Instytut Kardiologii, Warsaw
  - Woskowy Szpital Kliniczny, Wroclaw
- Hopitaux Universitaire de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided